CLINICAL TRIAL: NCT01482559
Title: Management of Hypotension In Preterm Infants: The HIP Trial Protocol for a Randomized Controlled Trial of Hypotension Management in the Extremely Low Gestational Age Newborn
Brief Title: Management of Hypotension In the Preterm Infant
Acronym: HIP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study ceased enrolling due to poor overall recruitment. Long-term follow up of enrolled participants ongoing.
Sponsor: University College Cork (Other)
Collaborators: Cork University Hospital (Other); Coombe Women and Infants University Hospital (Other); Royal College of Surgeons, Ireland (Other); National Maternity Hospital, Ireland (Other); University Hospital, Antwerp (Other); KU Leuven (Other); University of Alberta (Other); St. Justine's Hospital (Other); Institute for the Care of Mother and Child, Prague, Czech Republic (Other); GABO:mi (Industry); BrePco Biopharma Limited (Other); University College, London (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Clininfo S.A. (Industry)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Professor Eugene Dempsey, Consultant Neonatologist, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIP-FP7-BrePco; 2010-023988-17 (EudraCT Number)
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Hypotension; Low Blood Pressure; Intraventricular Hemorrhage of Prematurity
Keywords: Dopamine; Intraventricular haemorrhage; Periventricular Leukomalacia; Neurodisability; Infant
MeSH Terms: conditions — Hypotension; Leukomalacia, Periventricular | interventions — Dopamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dextrose 5% (Placebo Comparator): IV Infusion
  Interventions: Drug: Dextrose 5%
- Dopamine Hydrochloride (Experimental): IV Infusion
  Interventions: Drug: Dopamine hydrochloride

INTERVENTIONS:
Drug: Dopamine hydrochloride — Active drug substance 1.5 mg in 1 mL IV Infusion Minimum dose = 5mcg/kg/min Maximum dose = 20mcg/kg/min
  Other Names: ATC Code: C01CA04
  Arms: Dopamine Hydrochloride
Drug: Dextrose 5% — IV Infusion Minimum dose = 5mcg/kg/min Maximum dose = 20mcg/kg/min
  Other Names: Placebo
  Arms: dextrose 5%

SUMMARY:
The HIP trial is a large pragmatic, multinational, randomised trial of two different strategies for the management of hypotension in extremely low gestational age newborns (Standard with dopamine versus a restricted with placebo approach).

HYPOTHESIS: A restricted approach to the management of hypotension in extremely low gestational age newborns will result in improved neonatal and long-term developmental outcomes.

PRIMARY OBJECTIVE: To determine whether a restricted approach to the management of hypotension compared to using dopamine as first line pressor agent in infants born less than 28 weeks of gestation within the first 72 hrs after birth (transitional period), improves survival without significant brain injury at 36 weeks postmenstrual age (PMA) and improves survival without moderate or severe neurodevelopmental disability at 2 years corrected age.

DETAILED DESCRIPTION:
While hypotension - low blood pressure (BP) - is commonly diagnosed and treated in the very preterm infant there is enormous variation in clinical practice.Hypotension is statistically associated with adverse short-term and long-term outcomes however a systematic review of the literature was unable to find clear criteria to define hypotension. In addition the evidence to support current management strategies is minimal and mostly dependent on small studies that have measured short-term physiologic endpoints. Preterm infants who are diagnosed with and treated for low BP often have no biochemical or clinical signs of shock, they may have normal systemic blood flow, low systemic vascular resistance, and adequate tissue oxygen delivery and probably do not require treatment. Careful observation of such infants without intervention approach previously coined "permissive hypotension" may well be appropriate.

Excessive intervention in preterm infants may be unnecessary or even harmful. Analysis of a large neonatal database (Canadian Neonatal Network, CNN) demonstrated that treatment of hypotension was associated with an increase in serious brain injury. This remained true even after mean BP was included in the regression model suggesting that it may be the treatment of hypotension rather than the presence of hypotension which is harmful. The most common approach to treatment is to give one or more fluid boluses followed by dopamine. However, observational data have shown an association of fluid bolus administration with intracranial bleeding and in animal models correction of hypotension by rapid volume infusion can result in intraventricular haemorrhage; a complication which is associated with increased rates of death and neurosensory impairment in preterm human infants. Fluctuations in BP following commencement of inotropes are well recognised and could also trigger intraventricular haemorrhage. Furthermore dopamine the most commonly used inotrope has effects on many physiologic functions including pituitary effects which lead to secondary hypothyroidism a known risk factor for poor long-term neurodevelopmental outcome in the preterm infant. In addition dopamine elevates BP in the newborn predominantly due to vasoconstriction, which may be associated with a reduction in systemic perfusion.

There is no consensus on definitions of hypotension in the preterm infant. Many clinicians rely on absolute BP values alone to guide intervention. BP reference ranges are often based on birth weight, gestational age and postnatal age criteria. These statistically determined values vary considerably being based on observations of BP made in small cohorts of infants the majority of whom were born before the widespread implementation of important perinatal interventions (e.g antenatal glucocorticoid therapy) which are known to improve outcome and reduce the incidence of intraventricular haemorrhage in preterm infants. The Joint Working Group of the British Association of Perinatal Medicine has recommended that the mean arterial BP in mmHg should be maintained above the gestational age in weeks (e.g. an infant born at 25 weeks gestation should have a mean BP > 25mmHg). Despite little published evidence to support this 'rule', it remains the most common criterion used to define hypotension and it has been used in a number of recent randomised therapeutic intervention trials where it was the sole entry criteria. However, Cunningham et al have shown a poor relationship between this criterion and the incidence of intraventricular haemorrhage in preterm infants. In a separate study, the CNN report that 52% of preterm infants with birth weight < 1500g have a mean arterial BP less than their gestational age on the first day of life and thus may be diagnosed with and treated for hypotension.

It is uncertain whether hypotension (however defined) results in adverse clinical outcomes including adverse short-term outcomes (increased incidence of intraventricular haemorrhage) and adverse long-term neurodevelopmental outcome. Furthermore it is unclear whether intervention to treat hypotension results in improved outcomes. Dopamine is the most commonly used agent, an endogenous catecholamine that causes vasoconstriction and elevates BP, but has not been shown to improve clinical outcomes. Epinephrine is another endogenous catecholamine, which at low to moderate doses causes vasodilatation and stimulates cardiac function. It may increase perfusion when used in hypotensive neonates but the data are limited.

Current standard approaches to evaluation and treatment of transitional circulatory problems in the preterm infant are not evidence based. It is essential that these approaches be adequately investigated in this at risk group of infants.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age at birth less than 28 completed weeks, i.e. up to and including 27 weeks and 6 days.
2. Within 72 hours of birth
3. An indwelling arterial line, either umbilical or peripheral (e.g. radial, posterior tibial), suitably calibrated and zeroed, to monitor BP with the measuring dome at the level of the infant's mid-axillary line when supine
4. A pre-trial cerebral ultrasound scan demonstrating no evidence of grade 3 or 4 haemorrhage intraventricular haemorrhage (IVH)(i.e. intraparenchymal echodensity or echolucency, with or without acquired cerebral ventriculomegaly)
5. A mean blood pressure 1 mmHg or more below a mean BP value equivalent to the gestational age in completed weeks, which persists over a 15 minute period (mean BP < gestational age)

Exclusion Criteria:

1. Considered non-viable by attending clinicians.
2. Life-threatening congenital abnormalities including congenital heart disease (excluding patent ductus arteriosus, small atrial and/or ventricular septal defect). Infants known to require surgical treatment e.g. congenital diaphragmatic hernia, trache-oesophageal fistula, omphalocele, gastroschisis. Neuromuscular disorders. Frank hypovolaemia. Hydrops Fetalis.
3. Cranial ultrasound abnormality grade 3 IVH or more prior to enrolment

Ages: 23 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
First Co-Primary Outcome Measure: Survival to 36 weeks postmenstrual age free of severe brain injury | 36 weeks
  Survival to 36 weeks postmenstrual age free of severe brain injury (moderate or severe ventricular dilatation, intracerebral echodense lesions, and cystic periventricular leukomalacia) on cranial ultrasound at 36 weeks or discharge home which ever is the earlier.
Second Co-Primary Outcome Measure: Survival without moderate or serious disability as defined using consensus criteria for neurodevelopmental impairment. | 2 years of age
  Families will be offered routine appointments as per the local follow-up system. At 12-months, the physician will complete a simple disability assessment and all surviving infants will have a locally performed formal neurodisability assessment at 24 months age corrected for weeks of prematurity defined using criteria set out in the consensus statement "Health status...." (ww bapm.org/publications).

SECONDARY OUTCOMES:
All cause mortality at 36 weeks gestational age | 36 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Dempsey, Study Director — University College Cork; Peter Filan, Principal Investigator — Cork University Maternity Hospital; Gunnar Naulaers, Principal Investigator — KU Leuven; Zybnek Stranak, Principal Investigator — Univerzita Karlova v Praze; Keith Barrington, Principal Investigator — St. Justine's Hospital; Colm O Donnell, Principal Investigator — University College Dublin; Jan Miletin, Principal Investigator — Coombe Women and Infants University Hospital; Po-Yin Cheung, Principal Investigator — University of Alberta; David Corcoran, Principal Investigator — Royal College of Surgeons in Ireland; Neil Marlow, Principal Investigator — University College, London; Gerard Pons, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; David Van Laere, Principal Investigator — Neonatale Intensieve Zorgen; David Millar, Principal Investigator — Royal Maternity Hospital
Locations (10):
- Belgium (2):
  - University Hospital Antwerp, Antwerp, Edegem
  - Katholieke Universiteit Leuven, Oude God, Leuven
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
- Univerzita Karlova v Praze, Prague, Czechia
- Ireland (4):
  - Coombe Women and Infants University Hospital, Dublin, Dublin
  - Cork University Maternity Hospital, Cork
  - Royal College of Surgeons in Ireland, Dublin
  - University College Dublin, Dublin
- Royal Maternity Hospital, Belfast, United Kingdom

REFERENCES:
- [Derived] Dempsey EM, Barrington KJ, Marlow N, O'Donnell CPF, Miletin J, Naulaers G, Cheung PY, Corcoran JD, El-Khuffash AF, Boylan GB, Livingstone V, Pons G, Macko J, Van Laere D, Wiedermannova H, Stranak Z; HIP consortium. Hypotension in Preterm Infants (HIP) randomised trial. Arch Dis Child Fetal Neonatal Ed. 2021 Jul;106(4):398-403. doi: 10.1136/archdischild-2020-320241. Epub 2021 Feb 24. PMID 33627329